CLINICAL TRIAL: NCT03003845
Title: Activation of the Sphingosine-1-phosphate (S1P) to S1P1 Receptor Subtype (S1PR1) Axis in Patients With Interstitial Cystitis (IC) Pain : Identification of Potential Relevant Biomarkers
Brief Title: S1P1 Receptor Subtype (S1PR1) Axis in Patients With Interstitial Cystitis (IC) Pain
Acronym: S1P1
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Eugen C. Campian, MD, Principal Investigator, St. Louis University
Other Study IDs: 27338
Record Dates: First submitted 2016-11-22; First posted 2016-12-28 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — PERIPHERAL BLOOD LEUKOCYTE (PBLS) ANALYSIS (Research Related):
  Using immunoblotting, we will determine if the level of S1PR1 expression in peripheral blood leukocytes (PBLs) is increased in patients with IC pain. Patients will have blood samples taken, at the visit they sign the consent form 3 and 6 months later. A total of 4 teaspoons of blood will be taken for the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interstitial Cystitis: Patients with Interstitial Cystitis will be followed with Questionnaires and blood collection at 3, 6,and 12 months
  Interventions: Other: Questionnaires; Other: Collection of Blood samples

INTERVENTIONS:
Other: Questionnaires — QOL and pain questionnaires will be given to patients at 3, 6, and 12 months post surgery
Other: Collection of Blood samples — Blood for PBLs will be collected at 3, 6, and 12 months post surgery

SUMMARY:
For each patient in the study, blood, and pain scores will be collected to look for markers for pain, at the start of treatment and 6 months after surgery of treatment.

DETAILED DESCRIPTION:
The study is investigator-initiated, prospective, study. There will be no change in care.

Patients who have had a diagnosis of IC made by cystoscopy and hydrodistension and still have pain will be recruited for this study.

Patients will have blood samples taken at the visit they sign the consent form and 6 months later.

The study staff will call and remind the patient of their 6 month visit.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Patients must be able to provide written informed consent.
* Diagnosis of Interstitial Cystitis documented by provider

Exclusion Criteria:

* age <18 or >70 years of age
* pregnant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women are included. The onset of interstitial cystitis usually occurs between 30 and 70 years of age, with a median age of 43.
  .
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Visual Analog Scale at 6 months | 3 months
  S1PR1 levels in PBLs can discriminate patients with Interstitial Cystitis pain and patients with other types of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Eugen C Campian, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University Department of Obstetrics, Gynecology, and Women's Health, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No